CLINICAL TRIAL: NCT06951464
Title: A Phase II Study to Evaluate the Safety and Efficacy of Neoadjuvant Therapy With BL-B01D1 in Combination With Almonertinib Followed by Adjuvant Almonertinib in Patients With Epidermal Growth Factor Receptor Mutation Positive Stage II-IIIB Resectable Non-Small Cell Lung Cancer
Brief Title: A Study of BL-B01D1 and Almonertinib in Patients With Resectable EGFR+ Stage II-IIIB NSCLC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sichuan University (Other)
Responsible Party: Principal Investigator, Yongsheng Wang, Professor, Sichuan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BL-B01D1-206
Record Dates: First submitted 2025-04-23; First posted 2025-04-30 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — aumolertinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BL-B01D1 plus Almonertinib (Experimental): Neoadjuvant BL-B01D1 2.2 or 2.5mg/kg D1D8 Q3W plus Almonertinib 100mg QD
  Interventions: Drug: BL-B01D1; Drug: Almonertinib

INTERVENTIONS:
Drug: BL-B01D1 — BL-B01D1 (2.2 or 2.5mg/kg) to be administered on Day 1 and Day 8 of every 3-week cycle for 2 cycles.
Drug: Almonertinib — Almonertinib 100mg QD

SUMMARY:
This is a Phase II, open-labeled, single-arm, study of neoadjuvant BL-B01D1in combination with Almonertinib followed by adjuvant Almonertinib for the treatment of Patients with EGFR-Mutation Positive Stage II-IIIB Resectable Non-Small Cell Lung Cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily sign the informed consent form and comply with the study protocol requirements.
2. Male or female, Age ≥18 years and ≤75 years at the time of signing the informed consent form.
3. Diagnosed with stage II-IIIB (according to Version 8 of TNM staging) EGFR-sensitive mutation-positive non-small cell lung cancer (NSCLC) with feasibility or potential feasibility for radical surgery (radical lobectomy + systematic lymph node dissection), and assessed by the investigator as requiring neoadjuvant therapy.
4. Adequate pulmonary function to tolerate surgery.
5. Must have at least one measurable lesion per RECIST v1.1 criteria.
6. Eastern Cooperative Oncology Group (ECOG) performance status score of ≤1.
7. No severe cardiac dysfunction, with left ventricular ejection fraction (LVEF) ≥50%.
8. Organ function levels must meet the following criteria:

   1. Bone marrow function: Absolute neutrophil count (ANC) ≥1.5×10⁹/L, platelet count ≥100×10⁹/L, hemoglobin ≥90 g/L;
   2. Hepatic function: Total bilirubin (TBIL) ≤1.5×ULN, AST and ALT ≤2.5×ULN;
   3. Renal function: Serum creatinine (Cr) ≤1.5×ULN or creatinine clearance (Ccr) ≥50 mL/min (calculated by Cockcroft-Gault formula);
   4. Albumin ≥30 g/L.
9. Coagulation function: International normalized ratio (INR) ≤1.5 and activated partial thromboplastin time (APTT) ≤1.5×ULN.
10. Urine protein: ≤2+ on dipstick or ≤1000 mg/24h.
11. Contraception: Females of childbearing potential or males with partners of childbearing potential must use highly effective contraception from 7 days before the first dose until 6 months after the last dose. Females of childbearing potential must have a negative serum pregnancy test within 7 days prior to the first dose.

Exclusion Criteria:

1. Patients who have received previous systemic or local anti-tumor therapy for non-small-cell lung cancer.
2. Patients with other malignant tumors within 5 years before the first administration, except those who have been cured skin squamous cell carcinoma, basal cell carcinoma, superficial bladder cancer, prostate/cervix/breast cancer in situ and so on are considered to be eligible for enrollment.
3. Major surgery (investigator-defined) within 4 weeks before the first dose.
4. Current interstitial lung disease, drug-induced interstitial pneumonia, radiation pneumonitis requiring steroid therapy, or a history of these diseases.
5. Severe systemic infection occurred within 4 weeks before screening, including but not limited to severe pneumonia caused by fungi, bacteria, viruses, bacteremia, or serious infectious complications.
6. Patients at risk for active autoimmune disease, or with a history of autoimmune disease, Including but not limited to Crohn's disease, ulcerative colitis, systemic lupus erythematosus, sarcoidosis, Wegener syndrome, autoimmune hepatitis, systemic sclerosis, Hashimoto's thyroiditis, autoimmune vasculitis, autoimmune neuropathy (Guillain-Barre syndrome), etc. Exceptions include type I diabetes mellitus, hypothyroidism that is stable with hormone-replacement therapy (including that due to autoimmune thyroiditis), psoriasis or vitiligo that does not require systemic treatment, and hypothyroidism that is stable with hormone-replacement therapy.
7. Human immunodeficiency virus antibody (HIVAb) positive, active tuberculosis, active hepatitis B virus infection (HBsAg positive or HBcAb positive and HBV-DNA copy number > central detection lower limit) or hepatitis C virus infection (HCV antibody positive and HCV-RNA> central detection lower limit).
8. Poorly controlled hypertension (systolic blood pressure >150 mmHg or diastolic blood pressure >100 mmHg).
9. A history of severe cardiovascular and cerebrovascular diseases, including but not limited to:

   1. severe cardiac rhythm or conduction abnormalities, such as ventricular arrhythmia requiring clinical intervention, degree III atrioventricular block, complete left bundle branch block, frequent and uncontrollable arrhythmias, such as atrial fibrillation, atrial flutter, ventricular fibrillation, and ventricular flutter (except transient); h) prolonged QT interval (QTc>450 msec in men or QTc>470 msec in women) at rest (except transient);
   2. acute coronary syndrome, congestive heart failure, aortic dissection, stroke, or other grade 3 or higher cardiovascular or cerebrovascular event occurring within 6 months before the first dose;
   3. patients with New York Heart Association (NYHA) functional class ≥II heart failure;
   4. unstable angina pectoris;
   5. Patients with a history of cerebral infarction or cerebral hemorrhage within 6 months;
10. Previous history of allogeneic stem cell, bone marrow or organ transplantation.
11. Patients with a history of allergy to recombinant humanized antibodies or to BL-B01D1 or any excipients of Almonertinib Mesylate Tablets.
12. A history of autologous or allogeneic stem cell transplantation.
13. Pregnant or lactating women.
14. Other circumstances considered by the investigator to be inappropriate for participation in the trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-06-25 (Actual); Primary Completion 2027-05-05 (Estimated); Study Completion 2029-03-05 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response (pCR) | Approximately 9-11 weeks after the first dose
  Defined as absence of any viable cancer cells in the dissected tumour samples, including the main tumour, lymph nodes, and margins as assessed per central pathology laboratory post-surgery
Major Pathological Response (MPR) | Approximately 9-11 weeks after the first dose
  Defined as ≤10% residual cancer cells in the main tumour, as assessed per central pathology laboratory post-surgery

SECONDARY OUTCOMES:
Objective Response Rate（ORR） | Approximately 9-11 weeks after the first dose
  ORR is the proportion of subjects with CR or PR , based on RECIST v1.1.
Event-free survival (EFS) | From date of first administration up to approximately 5.5 years after the last patient is administrated
  An event is defined as documented disease progression that precludes surgery or prevents completion of definitive surgery; recurrence or a new lesion, local or distant (a new primary malignancy, confirmed by pathology if clinically feasible, is not considered to be an EFS event); death due to any cause
Disease free survival (DFS) | From date of first administration up to approximately 3.5 years after the last patient is administrated
  DFS is defined as the time from the date of surgery until the first date of disease recurrence (local or distant) or date of death due to any cause, whichever occurs first.
Overall Survival (OS) | From date of first administration up to approximately 5.5 years after the last patient is administrated
  OS will be defined as the time from the date of first dosing until death due to any cause
R0 resection rate | Approximately 9-11 weeks after the first dose
  R0 resection rate is defined as the proportion of subjects with complete surgical resection with microscopically negative margins (no residual cancer cells at the edges of the excised tissue).
The type, frequency and severity of adverse events during treatment (TEAE) and treatment-related adverse events (TRAE) | From the time of enrollment to either 28-days after the last dose of last study treatment for patients who do not undergo surgery, or 90-days post-surgery

OTHER OUTCOMES:
Biomarker expression in tumor tissues | From date of first administration up to approximately 5.5 years after the last patient is administrated

CONTACTS AND LOCATIONS:
Overall Officials: Yongsheng Wang, Principal Investigator — West China Hospital; Lunxu Liu, Principal Investigator — West China Hospital
Locations (1):
- West China Hospital, Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Chen Y, Mei J, Gao G, Zhang B, Li Y, Peng Z, Li C, Gan F, Pu Q, Liu C, Yang W, Liu L, Wang Y. A study protocol of a single-arm, prospective, open-label, non-controlled, phase II study of neoadjuvant BL-B01D1 combined with aumolertinib in resectable stage II-IIIB non-small cell lung cancer patients with EGFR mutation. Transl Lung Cancer Res. 2025 Dec 31;14(12):5527-5534. doi: 10.21037/tlcr-2025-829. Epub 2025 Dec 17. PMID 41510386